CLINICAL TRIAL: NCT05806086
Title: Clinical Effect of Panfoxol of Otolaryngological Diseases of Upper Respiratory Tract Infection: A Multicenter Retrospective Observational Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-087-01
Record Dates: First submitted 2023-02-20; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-02

CONDITIONS: Otologic Disease
Keywords: Panfoxol; Otologic Disease; Curative Effect; Upper Respiratory Tract Infection (URTI)
MeSH Terms: conditions — Ear Diseases; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Panfoshu + conventional treatment group（program-A） (Experimental): Panfoshu is commonly known as the product of bacterial dissolution. it was taken orally once a day on an empty stomach, one capsule at a time. 1 course of treatment was 6mon, which was taken 10 days a month, stopped for 20 days for 3 months, and observed for another 3 months(unmedicated). Usage and dosage: adults and adolescents above 12yrs take one capsule (7.0mg) every day, children (1yrs-12yrs) take one capsule (3.5mg) every day.
  Interventions: Drug: Panfoshu+Conventional Treatment（program-A）
- Panfoshu + conventional treatment group（program-B） (Experimental): Panfoshu was taken for 30 days in the first month, stopped in the second month, taken for 10 days and stopped for 20 days in a row for 3 months, and finally observed for 1 month. Usage and dosage: adults and adolescents above 12yrs take one capsule (7.0mg) every day, children (1yrs-12yrs) take one capsule (3.5mg) every day.
  Interventions: Drug: Panfoshu+Conventional Treatment（program-B）
- conventional treatment group (Other): Conventional medications are used to treat the relavant ear and nose symptoms.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Drug: Panfoshu+Conventional Treatment（program-A） — On the basis of conventional treatment, panfoshu combined therapy was added.Panfoshu was taken orally once a day on an empty stomach, one capsule at a time. 1 course of treatment was 6mon, which was taken 10 days a month, stopped for 20 days for 3 months, and observed for another 3 months(unmedicated). Usage and dosage: adults and adolescents above 12yrs take one capsule (7.0mg) every day, children (1yrs-12yrs) take one capsule (3.5mg) every day.
  Other Names: Bacteriolysis product
  Arms: Panfoshu + conventional treatment group（program-A）
Drug: Panfoshu+Conventional Treatment（program-B） — On the basis of conventional treatment, panfoshu combined therapy was added.Panfoshu was taken for 30 days in the first month, stopped in the second month, taken for 10 days and stopped for 20 days in a row for 3 months, and finally observed for 1 month. Usage and dosage: adults and adolescents above 12yrs take one capsule (7.0mg) every day, children (1yrs-12yrs) take one capsule (3.5mg) every day.
  Other Names: Bacteriolysis product
  Arms: Panfoshu + conventional treatment group（program-B）
Other: Conventional Treatment — Patients in this group were treated with only the conventional treatment.
  Arms: conventional treatment group

SUMMARY:
Patients with otolaryngological diseases caused by upper respiratory tract infections, including allergic rhinitis, chronic rhinosinusitis, secretory otitis media, and oblate gland hypertrophy, were treated with all drugs from Sun Yat-sen Memorial Hospital of Sun Yat-sen University, the First Affiliated Hospital of Sun Yat-sen University, Guangdong Provincial People's Hospital, and Guangdong Provincial Hospital of Traditional Chinese Medicine from January 2021 to December 2022. According to the treatment methods, the patients were divided into panfosol + conventional treatment group and conventional treatment group for multicenter retrospective analysis.

DETAILED DESCRIPTION:
FIrstly, Data of all patients were collected before and after treatment, including nasal endoscopy Lund Kennedy score, VAS scale for nasal/facial/olfactory symptoms, and ear/nose/snoring VAS scale, etc. According to the change values before and after treatment, the treatment results were divided into cure (complete control of the disease), effective (partial control of the disease), ineffective (uncontrolled disease). secondly, All participants were reviewed for gastrointestinal disturbances (nausea, abdominal pain, vomiting), skin reactions (rash, urticaria), respiratory discomfort (cough, dyspnea, asthma), and common problems (fever, fatigue, allergic reactions) after medication.

ELIGIBILITY:
Inclusion Criteria:

1. those who were diagnosed as ear, nose and throat diseases caused by upper respiratory tract infection, such as allergic rhinitis, chronic rhinosinusitis, secretory otitis media, and oblate gland hypertrophy
2. Complete clinical data were available at least once both before and after treatment

Exclusion Criteria:

1. Patients who are allergic to the ingredient panfosol
2. Autoimmune disease
3. Acute intestinal infection
4. Children younger than 1 year old
5. Patients diagnosed with nasopharyngeal carcinoma and other space-occupying diseases by imaging examination
6. Basic information is incomplete

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Therapeutic effective rate | through study completion, an average of 6 months.
  Treatment outcomes were classified as cure, effective, ineffective and relapse according to the condition after treatment. A cure means that the disease is under complete control, meaning that the patient's symptoms disappear completely and no medication is needed to continue treatment. Effective represents partial control of the disease, in which the patient's symptoms improve significantly but still require medication. Ineffective means the disease is not controlled or the symptoms are aggravated. Effective patients have symptoms aggravated, and the recurrence of symptoms after cure is defined as relapse.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | through study completion, an average of 6 months
  All participants were reviewed for gastrointestinal disturbances (nausea, abdominal pain, vomiting), skin reactions (rash, urticaria), respiratory discomfort (cough, dyspnea, asthma), and common problems (fever, fatigue, allergic reactions) after medication. Count the number of patients with these adverse symtoms.
Types, occurence rate and duration of the treatment-related adverse events | through study completion, an average of 6 months.
  All participants were reviewed for gastrointestinal disturbances (nausea, abdominal pain, vomiting), skin reactions (rash, urticaria), respiratory discomfort (cough, dyspnea, asthma), and common problems (fever, fatigue, allergic reactions) after medication. The presentation and duration of adverse symptoms in patients were counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China